CLINICAL TRIAL: NCT03362164
Title: Prospective Monocentric Cohort Study to Evaluate Predictors for Heart Failure and Sudden Cardiac Death in Patients With Fabry Disease
Brief Title: Evaluation of HEArt invoLvement in Patients With FABRY Disease
Acronym: HEAL-FABRY
Status: Recruiting | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Competence Network Heart Failure (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); St George's, University of London (Other)
Responsible Party: Principal Investigator, PD Dr. Peter Nordbeck, Head Consultant Cardiology and Chief of Electrophysiology, Wuerzburg University Hospital
Other Study IDs: FAZiT-2001
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Rare Diseases; Fabry Disease; Fabry Disease, Cardiac Variant; Hypertrophic Cardiomyopathy
Keywords: Fabry; Fibrosis; Dialysis; Stroke; Chronic kidney disease
MeSH Terms: conditions — Rare Diseases; Fabry Disease; Fabry Disease, Cardiac Variant; Cardiomyopathy, Hypertrophic; Fibrosis; Stroke; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ECG, Holter ECG, Echo, Cardiac MRI, Endomyocardial Biopsy, Kidney Biopsy, Cranial MRI, Skin Biopsy, EDTA Blood, Serum, Plasma, Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates predictors for the incidence of arrhythmias and sudden cardiac death as well as terminal heart failure in patients with Fabry disease.

DETAILED DESCRIPTION:
Fabry disease is a rare disease and part of the group of lysosomal storage disorders. Natural history of Fabry disease has proven poor survival to ages >50 years outlining the importance to evaluate cardiac symptoms and outcomes of patients with Fabry disease.

This study is a prospective cohort study and observes patients since 2001. Through this long-term experience and the relative high number of patients this study is suggested to help estimating the risk of cardiac arrhythmias and sudden cardiac death (SCD) as well as death or heart transplantation due to terminal heart failure.

All patients in treatment in the Fabry Center Wuerzburg (FAZiT) are included in this study if informed consent is provided.

ELIGIBILITY:
Inclusion Criteria:

* Fabry disease (genetically confirmed)
* Signed informed consent
* 18 years and older

Exclusion Criteria:

* No informed consent
* Withdrawal of informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes every patient with Fabry disease who is seen in the FAZiT Wuerzburg. No limitations are made.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2001-01 (Actual); Primary Completion 2032-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Cardiac death | From date of inclusion until the date of first documented event, up to the year 2032
  Patients sustaining cardiac death

SECONDARY OUTCOMES:
Heart transplantation | From date of inclusion until the date of first documented event, up to the year 2032
  On the basis of severe cardiac damage heart transplantation is needed
Malign Arrhythmias | From date of inclusion until the date of death, up to the year 2032
  Patients suffering any malign arrhythmias

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nordbeck, MD, PhD, Principal Investigator — Wuerzburg University Hospital
Locations (1):
- Wuerzburg University Hospital, Würzburg, Bavaria, Germany

REFERENCES:
- [Result] Oder D, Uceyler N, Liu D, Hu K, Petritsch B, Sommer C, Ertl G, Wanner C, Nordbeck P. Organ manifestations and long-term outcome of Fabry disease in patients with the GLA haplotype D313Y. BMJ Open. 2016 Apr 8;6(4):e010422. doi: 10.1136/bmjopen-2015-010422. PMID 27059467
- [Result] Seydelmann N, Liu D, Kramer J, Drechsler C, Hu K, Nordbeck P, Schneider A, Stork S, Bijnens B, Ertl G, Wanner C, Weidemann F. High-Sensitivity Troponin: A Clinical Blood Biomarker for Staging Cardiomyopathy in Fabry Disease. J Am Heart Assoc. 2016 May 31;5(6):e002839. doi: 10.1161/JAHA.115.002839. PMID 27247331
- [Result] Weidemann F, Maier SK, Stork S, Brunner T, Liu D, Hu K, Seydelmann N, Schneider A, Becher J, Canan-Kuhl S, Blaschke D, Bijnens B, Ertl G, Wanner C, Nordbeck P. Usefulness of an Implantable Loop Recorder to Detect Clinically Relevant Arrhythmias in Patients With Advanced Fabry Cardiomyopathy. Am J Cardiol. 2016 Jul 15;118(2):264-74. doi: 10.1016/j.amjcard.2016.04.033. Epub 2016 May 5. PMID 27265676
- [Result] Lenders M, Oder D, Nowak A, Canaan-Kuhl S, Arash-Kaps L, Drechsler C, Schmitz B, Nordbeck P, Hennermann JB, Kampmann C, Reuter S, Brand SM, Wanner C, Brand E. Impact of immunosuppressive therapy on therapy-neutralizing antibodies in transplanted patients with Fabry disease. J Intern Med. 2017 Sep;282(3):241-253. doi: 10.1111/joim.12647. Epub 2017 Jul 26. PMID 28682471
- [Result] Oder D, Liu D, Hu K, Uceyler N, Salinger T, Muntze J, Lorenz K, Kandolf R, Grone HJ, Sommer C, Ertl G, Wanner C, Nordbeck P. alpha-Galactosidase A Genotype N215S Induces a Specific Cardiac Variant of Fabry Disease. Circ Cardiovasc Genet. 2017 Oct;10(5):e001691. doi: 10.1161/CIRCGENETICS.116.001691. PMID 29018006
- [Result] Koping M, Shehata-Dieler W, Cebulla M, Rak K, Oder D, Muntze J, Nordbeck P, Wanner C, Hagen R, Schraven S. Cardiac and renal dysfunction is associated with progressive hearing loss in patients with Fabry disease. PLoS One. 2017 Nov 21;12(11):e0188103. doi: 10.1371/journal.pone.0188103. eCollection 2017. PMID 29161295
- [Derived] Lau K, Uceyler N, Cairns T, Lorenz L, Sommer C, Schindehutte M, Amann K, Wanner C, Nordbeck P. Gene variants of unknown significance in Fabry disease: Clinical characteristics of c.376A>G (p.Ser126Gly). Mol Genet Genomic Med. 2022 May;10(5):e1912. doi: 10.1002/mgg3.1912. Epub 2022 Feb 25. PMID 35212486
- [Derived] Liu D, Oder D, Salinger T, Hu K, Muntze J, Weidemann F, Herrmann S, Ertl G, Wanner C, Frantz S, Stork S, Nordbeck P. Association and diagnostic utility of diastolic dysfunction and myocardial fibrosis in patients with Fabry disease. Open Heart. 2018 Jul 12;5(2):e000803. doi: 10.1136/openhrt-2018-000803. eCollection 2018. PMID 30018776
- [Derived] Liu D, Hu K, Schmidt M, Muntze J, Maniuc O, Gensler D, Oder D, Salinger T, Weidemann F, Ertl G, Frantz S, Wanner C, Nordbeck P. Value of the CHA2DS2-VASc score and Fabry-specific score for predicting new-onset or recurrent stroke/TIA in Fabry disease patients without atrial fibrillation. Clin Res Cardiol. 2018 Dec;107(12):1111-1121. doi: 10.1007/s00392-018-1285-4. Epub 2018 May 24. PMID 29797054